CLINICAL TRIAL: NCT01855906
Title: The Impact of Total Knee Arthroplasty Surgical Technique on Coronal Plane Motion and PatelloFemoral Articulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103307
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Total knee replacement; Gap balanced; Measured resection
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gap balanced surgical technique (Active Comparator): Study patients in this arm of the study will have their knee replacement done using the gap balanced technique. Gap balancing adjusts the bony cuts for femoral rotation to balance the soft tissues of the knee in flexion.
  Interventions: Procedure: Gap balanced surgical technique
- Measured resection surgical technique (Active Comparator): Study patients in this arm of the study will have their knee replacement done using the measured resection surgical technique. Pre-determined bony cuts are made and appropriate balance is obtained by judicious soft tissue releases as required.
  Interventions: Procedure: Measured resection

INTERVENTIONS:
Procedure: Gap balanced surgical technique — Gap balanced surgical technique
  Arms: Gap balanced surgical technique
Procedure: Measured resection — Measured resection surgical technique
  Arms: Measured resection surgical technique

SUMMARY:
The purpose of this study is to examine the impact of two surgical techniques on the outcome of the knee replacement surgery.

DETAILED DESCRIPTION:
How stable a total knee replacement is depends on the correct and precise rotation of the femoral component. Abnormal femoral component rotation has been associated with numerous adverse conditions including knee instability, knee pain, scar tissue, and abnormal knee motion. Controversy exists, however, regarding the most favorable surgical technique to determine accurate femoral component rotation. Some doctors prefer a measured resection technique in which landmarks on the femur bone are used to determine where to place the femoral component. Others recommend a gap-balancing technique in which the femoral component is positioned by balancing the ligaments of the knee and placing it in the position where each ligament is equally strained.

The purpose of this study is to examine the impact of the measured resection and gap-balancing surgical technique on how the total knee replacement moves and patient knee outcome scores. Knee outcome scores are assessed from the responses given by patients to questions about outcomes associated with total knee replacement related to pain, symptoms, activities of daily living, sport and recreational function, and knee-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon and patient have determined that patient requires a primary total knee arthroplasty and agrees to participate and signs the informed consent for study.

Exclusion Criteria:

* History of alcoholism
* Unable to speak English
* Inflammatory Arthritis
* Pregnant women or any woman with plans to begin a family.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective will be to assess coronal balance through a range of motion. | One year post-operatively
  Assessed through dynamic fluoroscopic analysis.

SECONDARY OUTCOMES:
Patellofemoral tracking | One year post-operatively
  Assessed using dynamic fluoroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD., Principal Investigator — London Health Sciences Centre - University Hospital
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada